CLINICAL TRIAL: NCT06638723
Title: Enhancing Motor Function in Individuals with Lower Limb Amputation Through Peer-Based Balance and Fall Recovery Skill Training
Brief Title: Enhancing Motor Function in Individuals with Lower Limb Amputation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UNLV-2022-99; W81XWH-22-1-0216 (Other Grant/Funding Number: Department of Defense (CDMRP))
Record Dates: First submitted 2023-11-27; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Amputation
Keywords: limb loss; peer support; motor learning; EEG; falls; balance; prosthetics

STUDY DESIGN:
Intervention Model Description: The same group of participants will experience the two conditions, separated by a 4-week washout period. The initial condition is randomly decided.
Who Masked: Participant
Masking Description: Participants were randomized to experience one of the two conditions (amputee peers vs. non-amputees) demonstrating how to perform motor tasks. Participants were masked to the study hypothesis and the existence of the other group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amputee peers (Experimental): This research uses a cross-over design to expose the participants with lower limb loss to the two training conditions (observing amputee peers vs. non-amputees) in random order, with a 4-week washout period between conditions. In this arm, participants are instructed to learn from video demonstrations by amputee peers. The videos will show balance and fall recovery movement tasks performed by the models, 15-30 seconds in length. The instruction to the participants is: "Please watch and learn the tasks as performed by the demonstrator. You (the participant) will be asked to perform these tasks later."
  Interventions: Behavioral: Balance and fall recovery training
- Non-amputees (Experimental): In this arm, participants with lower limb loss are instructed to learn from video demonstrations by non-amputees. The videos will show balance and fall recovery movement tasks performed by the models, 15-30 seconds in length. The instruction to the participants is: "Please watch and learn the tasks as performed by the demonstrator. You (the participant) will be asked to perform these tasks later."
  Interventions: Behavioral: Balance and fall recovery training

INTERVENTIONS:
Behavioral: Balance and fall recovery training — Following the video observation described in the arms, participants will undergo training to physically practice the motor tasks. The training will take place over a 2-week period encompassing 40 practice trials for each task over the training sessions. During training, the investigators will continuously monitor the changes in balance and fall recovery task performance, and will provide feedback. Participants can request to re-watch the demonstration video that they were assigned to at any time.

SUMMARY:
The overall goal of this research project is to investigate the effectiveness and the science of peer-based prosthetic skill training in individuals with leg amputation. Our belief is that amputee learners will show improved skill learning when observing demonstrations from other amputees, as opposed to observing nonamputee models. The investigators will accomplish the objective by answering the following two questions:

Question 1: Does peer-based observation training works better for learning motor tasks for individuals with lower limb amputation (LLA)?

Question 2: Are there differences in visual focus, behavior, and brain activation patterns when observing motor task demonstrations from amputee peers vs. non-amputees?

Participants of this study will be asked to learn a balance and a fall recovery task by observing video demonstrations by amputee peers vs. non-amputees. The investigators will compare which setting produce better learning.

DETAILED DESCRIPTION:
Objective/Hypothesis: The overall objective of this project is to investigate the clinical scientific bases of peer observation sensori-motor skill training in individuals with lower limb amputation. The general hypothesis is that participants observing models who share the same levels of amputation with them (i.e. amputee peers) will exhibit traits of enhanced motor learning when compared to observing non-amputee models. Knowledge gained from this study will directly benefit the development of more effective rehabilitation protocols and has the potential to fundamentally transform the clinical practice of post-amputation rehabilitation.

Aim 1: Determine the effects of peer-based observation training on sensori-motor performance and learning in individuals with LLA. During a 2-week training period, the investigators will assess the differences in task performance and learning outcomes between participants who are instructed to learn to perform the tasks (i.e. balance and reactive fall arrest) by observing video demonstrations from amputee peers vs. non-amputees (n=20).

Aim 2: Examine the differences in visual focus, behavioral psychometrics, and brain activation patterns during and after observing motor task demonstrations from amputee peers vs. non-amputees. The investigators will compare the differences in visual focus time, task-specific self-efficacy, adopted mindset, and event-related brain activation patterns between the two conditions where participants learn to perform the motor tasks demonstrated by amputee peers vs. non-amputees.

Study Design: This research will use a cross-over design with a washout period to expose the participants to the two conditions in random order. In Aim 1, participants with unilateral LLA will be instructed to watch video demonstration of balance and fall recovery tasks performed by either an amputee peer or non-amputee with the intention of learning to perform the task. The subsequent 2-week training will consist of 60 practice trials for each task (over at least 3 sessions).

Participant's task performance (measured by time-in-balance during the balance task, and peak trunk flexion angle and rate of successful fall arrest during the fall recovery task) will be tracked before, throughout, and after (retention) training. To accomplish Aim 2, the investigators will evaluate and quantitatively measure the participant's visual focus (using eye tracking technology), psychometric traits (self-efficacy, motivation, and growth mindset), and brain activation patterns (assessed by electroencephalography, EEG) during the video observation and the corresponding training period.

ELIGIBILITY:
Inclusion Criteria:

* 1) have unilateral lower limb amputation,
* 2) age >18 years,
* 3) are properly fitted with a walking prosthesis and use it regularly with at least moderate proficiency (K-2 level or above, further defined as scoring greater than 50 percentile on the Prosthetic Limb Users Survey of Mobility),
* 4) able to stand for at least 5 minutes without using an assistive device or experiencing excessive fatigue,
* 5) willing to travel to UNLV 6 times for training and testing.

Exclusion Criteria:

* 1) have other concurrent central nervous system diseases that influence motor function and balance,
* 2) have leg/foot ulcer or other conditions that cause pain during weight-bearing,
* 3) have cardiovascular, respiratory or other critical health conditions that preclude moderate physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Balance performance | During the 6-visit training (3 months from the first to last visit)
  During balance training, a potentiometer and a timer integrated to the balance platform will monitor the sway angle of the platform and time-in-balance, which is defined as when the platform angle is within ± 5° of horizontal. The primary outcome measure is time in balance (seconds) during each 30-second balance trial.
Fall recovery performance (frequency) | During the 6-visit training (3 months from the first to last visit)
  During fall recovery training, the incidence of falls during the trials will be recorded
Fall recovery performance (movement quality) | During the 6-visit training (3 months from the first to last visit)
  During fall recovery training, the trunk and lower extremity stepping kinematics during the trials will be recorded
Patient's self-reported psychometric outcomes | During the 6-visit training (3 months from the first to last visit)
  Surveys will be used to assess the participant's perceptions about the training, task-specific self-efficacy, and learning mindset.
  Task-specific self-efficacy questions will be answered on an analog scale of 0-100 and included: "How difficult do you think the task is?", "How confident are you that you will be able to perform the task after practice?", and "How useful do you think this training is when applied to real life situations?".
  Growth mindset survey will ask the participants to rate a series of statements including: "I can always improve how well I conduct a physical task (such as maintaining balance or walking).", "I only have a certain amount of physical capacity, and I can't really do much to change it.", "Hard work is needed to master skills needed for different tasks.", and "Other people's successes are inspiring. I can learn by their example."

SECONDARY OUTCOMES:
Visual focus assessment using eye tracking | During video observations at the beginning of the 6-visit training (1st and 4th visits). The training is 3-months long.
  During demonstration video-watching, monocular recordings of the participant's eye movements will be recorded simultaneously by a desktop mounted eye-tracker. The coded data will be used to compare the visual attentional focus between the amputee-peers vs. non-amputee videos.
Brain activation pattern assessment using electroencephalography (EEG) | During video observations at the beginning of the 6-visit training (1st and 4th visits). The training is 3-months long.
  During demonstration video-watching, participants' brain activity will be assessed using a non-invasive, battery-powered EEG recording system with 64 electrodes on their head.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Ping Lee, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
There is currently not a plan to share participant data with other researchers.

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Wulf G, Chiviacowsky S, Lewthwaite R. Altering mindset can enhance motor learning in older adults. Psychol Aging. 2012 Mar;27(1):14-21. doi: 10.1037/a0025718. Epub 2011 Oct 10. PMID 21988153
- [Background] Cusack WF, Thach S, Patterson R, Acker D, Kistenberg RS, Wheaton LA. Enhanced Neurobehavioral Outcomes of Action Observation Prosthesis Training. Neurorehabil Neural Repair. 2016 Jul;30(6):573-82. doi: 10.1177/1545968315606992. Epub 2015 Oct 5. PMID 26438442